CLINICAL TRIAL: NCT05547555
Title: IVF Outcomes Based on Invasive PGT-A Embryo Selection Versus Non Invasive PGT-A Assisted
Brief Title: Invasive PGT-A Embryo Selection Versus Non Invasive PGT-A Assisted Embryo Selection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assisting Nature (Other)
Responsible Party: Principal Investigator, Papanikolaou Evaggelos, MD, PhD, Fertility Specialist, Scientific Director at Assisting Nature IVF Clinic, Assisting Nature
Other Study IDs: AN010
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Infertility; Aneuploidy; Chromosome Abnormality
Keywords: IVF; PGT-A; NON- INVASIVE PGT-A; TIME LAPSE; EMBRYO SELECTION
MeSH Terms: conditions — Infertility; Aneuploidy; Chromosome Aberrations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- INVASIVE PGT-A: Women who proceed to embryo transfer after invasive PGT-A embryo selection.
  Interventions: Diagnostic Test: embryo selection
- NON INVASIVE PGT-A: Women who proceed to embryo transfer after non- invasive PGT-A embryo selection.
  Interventions: Diagnostic Test: embryo selection

INTERVENTIONS:
Diagnostic Test: embryo selection — The basis of embryo selection for transfer: invasive PGT-A or after non-invasive PGT-A

SUMMARY:
This is a prospective randomised study of the evaluation of the clinical IVF results after invasive PGT-A embryo selection versus Non-invasive PGT-A assisted embryo selection in subfertile women.

DETAILED DESCRIPTION:
A randomized prospective study focusing on subfertile women undergoing IVF treatment followed by embryo transfer on the blastocyst stage.

Women assigned to group A proceed to embryo transfer, after invasive PGT-A embryo selection, while women of group B after non-invasive PGT-A assisted embryo selection.

IVF outcomes, regarding the success rate of the trasnfer and the time required to achieve conception is studied in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Women who followed IVF treatment
* 40 years old or older
* Single embryo transfer
* blastocyst stage cultured embryos

Exclusion Criteria:

* women under the age of 40 years
* not blastocyst transfer (transfers performed at earlier embryo stage)
* double embryotransfer
* women who had embryotransfer according to morphological criteria women whose embryos were not time-lapse monitored

Ages: 40 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women 40 years old or older who were divided in two groups according to the embryo selection criteria for embryotransfer: women in group A proceeded to embryo transfer after invasive PGT-A assisted embryo selection and women in group B proceeded to embryo transfer after non- invasive PGT-A assisted embryo selection.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Embryotransfers to conceive | Up to the embryotransfer of the last enrolled patient (Dec 2023)
  The number of the embryotransfers required for women to conceive
Time interval to conceive | Up to the pregnancy test after the last embryo transfer of an enrolled patient (Jan 2024)
  Time interval required for women to conceive (in months): from day of first embryotransfer to positive hCG test
Cumulative Live Birth Rate | Up to 38 weeks after the embryo transfer
  Cumulative Live Birth Rate achieved after one OPU treatment

SECONDARY OUTCOMES:
Abortion rate | Up to 2nd trimester miscarriages
  The spontaneous miscarriage of women in both groups
DaC rate | during pregnancy according to Greek Law
  The rate of the dilation and curretage rate in both groups

CONTACTS AND LOCATIONS:
Locations (1):
- Assisting Nature, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided